CLINICAL TRIAL: NCT01351181
Title: A Case Control Study to Assess the Effectiveness of Written Advice to Increase Physical Activity Given to Type II Diabetics by Nursing Staff During the Diabetic Annual Review in UK General Practice
Brief Title: Physical Activity Advice in Diabetics at Annual Review
Acronym: PAADAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ship Street Surgery (Other)
Responsible Party: Dr J D HILL, Ship Street Surgery
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 007489
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise advice (Experimental): Behavioural
  Interventions: Behavioral: Leaflet; Behavioral: Exercise Advice
- Normal Care (Other): Normal care
  Interventions: Behavioral: Normal Care

INTERVENTIONS:
Behavioral: Leaflet — Advice Leaflet
  Arms: Exercise advice
Behavioral: Exercise Advice — Leaflet
  Arms: Exercise advice
Behavioral: Normal Care — Normal Care
  Arms: Normal Care

SUMMARY:
Type II diabetes is an important condition with a UK prevalence of 3.54% affecting approximately 2.5 million people across the country. Diabetics have a fivefold increased risk of cardiovascular disease and over 65% of diabetics will die from coronary heart disease or stroke. Exercise is one of the management tools along with medication and weight reduction available to improve diabetic control reducing morbidity and mortality. Exercise promotion might be more effective at a population level if it could be incorporated in a simple form as part of pre-existing routine care. This case control study seeks to assess the effectiveness of written exercise advice given to Type II diabetics at the time of their annual review. The study will be open to all Type II diabetics in a single general practice attending their routine nurse led annual review. The intervention uses leaflets prepared as part of a previous study the Time2Act study and assessment will be by self-reported questionnaires. Follow up will be over 12 months but the study design will allow for longer durations. Previous studies have demonstrated the effectiveness of exercise as an intervention but have often been hospital-based and used exercise interviews as the main intervention rather than incorporating exercise advice into structures already established in routine Primary Care. If this study demonstrates that a simple intervention carried out as part of routine care has a positive effect if only at a low level then disseminating this knowledge across the country would bring significant benefits to Type II diabetics.

DETAILED DESCRIPTION:
Study Objectives

The objectives of this study are to evaluate whether incorporating a simple low-cost, low resource intervention into routine diabetic care in General Practice is effective in producing a sustained change in activity levels across significant numbers of patients. Even if the change in activity level is small on an individual patient level but is widespread across the practice's diabetic population then the intervention will be of value. The primary outcome will be measured using a validated self reporting questionnaire (SPAQ-Scottish Physical Activity Questionnaire) to measure changes in the amount of exercise undertaken. During routine diabetic care a wide range of information is recorded on the clinical system in part to satisfy QoF (Quality and Outcomes Framework) requirements it will be possible to further analyse the dataset by parameters such as age, sex and social class as well as seeing whether there is a change in blood pressure, weight, lipid profile and HbA1C (glycosylated haemoglobin- a measure of medium term diabetic control). The intervention is simple and if effective could form part of the routine ongoing care of Type II Diabetics. If extended over a longer period it might be possible to extract data relating the intervention to illness and death rates.

The delivery of an intervention, from a known Health Care Professional in a familiar setting, at an interview where the patient's expectation is to receive advice and hopefully therefore be receptive to that advice, with regular reinforcement as part of routine care may mean that the initial intervention can be straight forward. This study seeks to answer this question by deliberately choosing written information which was in an unsuccessful arm of a previous study ~ the Time2Act study.

The original study design was to record baseline activity levels in the target population with an appropriate assessment tool, carry the intervention and then record any changes in activity levels and biometric and biochemical parameters at intervals . This could have been considered as an audit and part of 'normal care' and therefore some investigators might argue that formal patient consent was not required. However following discussions with the team at Queen Mary's University of London (QMUL) this would weaken the study as it would be difficult to assess the effects of any confounding factors. The presence of a control group would make the study more valid. A randomized controlled trial (RCT) would have been the ideal design but constraints of time and outcomes measured by a questionnaire would have required a larger than practical study of long duration. A Case Control study was therefore chosen and will act as a pilot for follow up work.

Inclusion and Exclusion Criteria

All Type II diabetics over 18 attending the Diabetic Annual Review (DAR) will be eligible to be included in the research. The DAR is offered between 3 and 12 months from initial diagnosis. This will exclude newly diagnosed diabetics who might have undergone DESMOND courses. Type II diabetics under 18 are followed up by the paediatric team and would not normally be called for review in the practice. Other exclusion criteria relate to conditions where the patient is either unable to understand the advice given or physically unable to follow it. Patients with dementia who are physically able to participate will not be excluded as long as consent can be obtained from them or their next of kin or legal representative. Input from their General Practitioner (GP) in the surgery will be valuable here.

Consent

Written consent will be sought from all participants. Consent will be obtained by the site investigator Dr J D Hill following a written invitation. They will be an opportunity for individuals to discuss the study face to face with Dr Hill or the registered GP. The GPs will have had information about the study in writing as well as discussed it at a Practice meeting.

The benefits of activity should be available to all diabetics and it is important that patients with limited understanding are not excluded. Consent would therefore be sought from their responsible carer e.g. someone who hold power of attorney or similar instrument. Pre-notification lists will be passed to the registered GP prior to invitations being sent out to allow them to exclude inappropriate patients e.g. terminally ill. The main researcher has experience in assessing capacity in his full time work as a General Practitioner.

Risks, Burdens and Benefits

To a degree there is some risk to participants in both arms of the study. The intervention group who will be encouraged to increase their activity levels could be construed to be at risk from injury from unaccustomed exertion (e.g. muscle aches) or it may reveal an underlying undiagnosed pathology (e.g. angina). The advice leaflet has been carefully designed to provide a graded increase in activity to minimize these risks and participants will have the opportunity as the study is based in their surgery to seek advice regarding any unexpected symptoms.

For the duration of the study the control group will receive 'normal care' in all respects including general advice to increase activity and access to information from Diabetes UK. They may perceive this as a lower level of care. Both groups will have increased contact with the surgery during the study which will be organized in such a way to minimize intrusion.

The benefits are expected in two phases. Initially the intervention group should see a positive health return on their increased activity which will then be rolled out as part of normal care across the whole patient population.

Confidentiality

Data handling within the surgery is subject to tight controls overseen by the nominated Caldicott guardian and the practice is compliant with the regulations attached to the IMT DES (Information Technology Direct Enhanced Service) which is regulated by West Sussex PCT. Information will be held on the secure Clinical System. Staff handling patient information will have access to this data as part of their normal duties and will be subject to NHS codes of confidentiality. For statistical analysis off site patients surgery number (not NHS number) will be used as an identifier. The only way to trace this back to an individual would be to have access to the password protected Surgery system. Information which comes to light during the study indicating a serious risk will be fed back to the main investigator and thence to the registered GP.

Investigator as General Practitioner

During the study period patient contacts will take place where it may be clinically appropriate to encourage exercise to a study participant. One's primary responsibility is for patient care independent of the study so advice will not be withheld but any written information given will be from organizations such as Diabetes UK and not the study leaflet. Normal care will therefore be maintained. At the end of the study future practice will be guided by the results.

ELIGIBILITY:
Inclusion Criteria:

* Adult Type 2 diabetics

Exclusion Criteria:

* non ambulatory
* within 6 months diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
SPAQ score | 12 months
  Increased Physical Activity

CONTACTS AND LOCATIONS:
Overall Officials: Jerry D Hill, MRCGP, Principal Investigator — National Health Service, United Kingdom
Locations (1):
- Ship Street Surgery, East Grinstead, Sussex, United Kingdom